CLINICAL TRIAL: NCT06946563
Title: Fetoscopic Neural Tube Defect Repair: Observational Pilot Study
Brief Title: Fetoscopic Neural Tube Defect Repair
Acronym: NTD
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Raphael Sun, Principal Investigator, Oregon Health and Science University
Other Study IDs: OHSU IRB 24397
Record Dates: First submitted 2025-03-18; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Neural Tube Defects; Spina Bifida
Keywords: Fetal Surgery; Fetoscopy
MeSH Terms: conditions — Neural Tube Defects; Spinal Dysraphism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Fetoscopic Neural Tube Defect Repair: Individuals who undergo fetoscopic Neural Tube Defect (NTD) repair. Participants will undergo fetal surgery between 24 weeks 0 days and 27 weeks 6 days.
  Interventions: Device: Fetoscopic Neural Tube Defect Repair Devices

INTERVENTIONS:
Device: Fetoscopic Neural Tube Defect Repair Devices — Fetoscopic NTD repair will be performed on enrolled participants. An incision will be made to gain exposure and access to the uterus. The amniotic cavity is entered using a needle to administer fetal anesthesia. Then, the initial trocar is inserted into the amniotic cavity. The major steps of the procedure are neural placode dissection, myofascial flaps creation, and closure of the neural tube defect.
  Other Names: Karl Storz Endoscopy-America, Inc.; Richard Wolf Medical Instruments, Corp.; Advanced Endoscopy Devices; Lexion Medical, LLC.; Cook Medical, Inc.; Becton Dickinson Visitec Pro; TERUMO Pinnacle; Integra LifeSciences; Applied Medical Resources

SUMMARY:
This is a single-arm prospective study to record maternal and neonatal outcomes on subjects who undergo fetoscopic repair of Neural Tube Defects (NTD) at Oregon Health & Science University (OHSU). Fetoscopic repair will take place between 24 weeks 0 days and 27 weeks 6 days gestation. Surgical, post-operative, delivery, and neonatal outcomes will be collected.

DETAILED DESCRIPTION:
Patients undergoing fetoscopic NTD repair will be enrolled. Possible surgical approaches include completely percutaneous, laparotomy assisted, or mini laparotomy. Surgical approach will be determined by placental location, maternal body habitus, and shared decision making with the patient. The actual fetoscopic NTD repair is the same regardless of the surgical approach. Follow-up data collection will occur post-operatively, at delivery, NICU admission, and throughout childhood.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 18 years or older
* Capable of consenting for their own participation in the study
* Decision to have fetoscopic repair following counseling of all options
* Open spina bifida with the upper boundary between T1 and S1
* Gestational age between 24 0/7 to 26 6/7 weeks' gestation at the time of surgery
* Normal karyotype and/or normal chromosomal microarray by invasive testing. In the case of a microdeletion, microduplication, or variant of uncertain significant, the decision to include or exclude will be at the discretion of the Principal Investigators.
* Absence of major cardiac anomalies confirmed by fetal echocardiogram
* Adequate social support throughout pregnancy
* Parental or guardian willingness to undergo follow-up evaluations of the child after birth

Exclusion Criteria:

* Multiple gestation
* Major fetal anomalies unrelated to the neural tube defect
* Kyphosis in fetus of 30 degrees or more as assessed by ultrasound or MRI
* Previous spontaneous singleton preterm birth prior to 37 weeks
* Presence of cervical cerclage at the time of surgery or history of cervical insufficiency
* Cervical length less than 20 mm by endovaginal ultrasound
* Placenta previa or evidence of placental abruption
* Technical factors such as large uterine fibroids, uterine anomalies, or fetal membrane separation for which the risks of surgery are deemed to outweigh the benefits
* Maternal obesity precluding surgical access with a BMI > 45 or if the Principal Investigator determines the body habitus to be technically challenging
* Alloimmunization in pregnancy including Kell sensitization or a history of neonatal alloimmune thrombocytopenia
* Maternal HIV or Hepatitis B positive status. If the patient's HIV or Hepatitis B status is unknown, the patient must be tested and found to be negative prior to surgery
* Known Hepatitis C positivity. If the patient's Hepatitis C status is known, they do not need to be screened
* Maternal medical condition which is a contraindication to surgery or general anesthesia. This includes previous hysterotomy in the active segment of the uterus
* Maternal medical co-morbidities which would significantly increase the risk of spontaneous or iatrogenic preterm delivery
* Inability of the patient to comply with travel and follow-up requirements of the study
* Patient not meeting psychosocial criteria determined by fetal care social worked to comply with the medical care and plan for follow ups
* Participation in another interventional study that influences maternal and fetal morbidity and mortality
* Known history of hypersensitivity to collagen products or chondroitin materials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant patients with a diagnosed Neural Tube Defect (NTD) electing to undergo fetoscopic NTD repair.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of minimally invasive surgical repair of NTD in fetus | At the time of NTD repair surgery
  Whether closure was achieved and whether the case was completed using the fetoscopic technique

SECONDARY OUTCOMES:
Chiari II malformation reversal | Post-surgery ultrasound (weekly from surgery to delivery), post-surgery fetal MRI (4-6 weeks after surgery), and postnatal MRI (5-7 days after birth)
  Reversal of hindbrain herniation based on ultrasound, fetal MRI, and postnatal MRI

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Sun, MD, Principal Investigator — Oregon Health and Science University; Andrew Chon, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States